CLINICAL TRIAL: NCT00764075
Title: CT and 3D-Echocardiography Placement of CRT-Leads
Brief Title: Guided Placement of CRT-Leads
Acronym: EK138/08
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Christian Knackstedt, MD, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRT-Study
Record Dates: First submitted 2008-09-26; First posted 2008-10-01 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure
Keywords: heart failure; EF<35%; NYHA II, III or IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): guided implantation of the left ventricular lead
  Interventions: Device: Beutel TM
- 2 (Placebo Comparator): standard implantation of the left ventricular lead
  Interventions: Other: standard
- Pilot Group (Experimental): feasibility of guided placement of CRT-leads in 20 Patients
  Interventions: Device: software Beutel TM

INTERVENTIONS:
Device: Beutel TM — application of BeutelTM
  Arms: 1
Other: standard — standard procedure will be applied but no Beutel TM software
  Arms: 2
Device: software Beutel TM — application of BeutelTM to patients data for determination of site of latest contraction
  Arms: Pilot Group

SUMMARY:
In this open, prospective, randomized, parallel group, German-American, two-center, Phase I study the standard-approach CRT-implantation will be compared to a guided CRT-implantation after determining the site of latest contraction and placement of the electrode as close as possible to this site, using a 5-step-scheme of imaging methods determining the site of latest contraction prior to implantation.

DETAILED DESCRIPTION:
Patients will be allocated to two groups with either

1. Guided implantation of the left ventricular lead
2. Empirical implantation of the left ventricular lead (current clinical standard)

For Treatment Group a) the target vessel, which is the vessel with smallest distance between RLC and CVS is determined in advance and provided to the implanting physician. In case, this vessel is not amenable for lead positioning, a second vessel which is the second closest to the RLC is defined.

For Treatment Group b), the physician has to choose the vessel where to place the electrode without knowing the exact spatial orientation between that particular side-branch and the RLC.

In all patients, standard biventricular devices and leads are to be used. Aspects that are evaluated are:

1. Technical success in placing the electrode in the target vessel.
2. Failure due to dislocation during the implantation procedure or phrenic nerve stimulation.

Also, procedure duration, radiation exposure, and complications occurring during the procedure as well as post- operatively will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure,
* Ejection fraction <35%,
* Complete left bundle branch block >120ms,
* NYHA II,III or IV

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria or not capable/mental able to understand and follow the instructions;
* Impaired kidney function (GFR <30ml/min;
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of non-responders regarding ejection fraction | 6 months

SECONDARY OUTCOMES:
rate of non-responders regarding NYHA-classification, left end-diastolic and end-systolic volume | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Knackstedt, MD, Principal Investigator — RWTH Aachen University Departement of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonology and Vascular Medicine, Aachen, North Rhine-Westphalia, Germany